CLINICAL TRIAL: NCT03624296
Title: Characterization of Cortical Injury in Early MS Patients: a 7T MRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-35; 2018-A00928-47 (Other: n°IDRCB)
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with multiple sclerosis (MS) (Experimental)
  Interventions: Device: MRI 7T; Other: TEST EDSS; Other: TEST MSFC

INTERVENTIONS:
Device: MRI 7T — MRI 7T
Other: TEST EDSS — EDSS - Expanded Disability Status Scale
Other: TEST MSFC — MSFC - Multiple Sclerosis Functional Composite

SUMMARY:
The main aim of the present study is to assess the prevalence, the topography and the clinical counterpart of cortical lesions in patient included early after the first clinical episode of multiple sclerosis. A second aim is to assess the direct contribution of cortical lesions - independent of WM injury - on the diffuse grey matter damage.

Thirty MS patients will be included in the six months after the first clinical episode of multiple sclerosis for a monocentric transversal MRI study at 7T to assess cortical MS injury. Clinical (EDSS) and neuropsychological assessments will be performed in the population the same day of a multi-parametric MRI. MRI protocol is designed to increase the detection rate of CL using multiple contrasts at high isotropic resolution (600µm3) on a whole brain exploration. Thus, MRI acquisition will include MP2RAGE, T2*, FLAIR and DIR as previously published but also recent MRI technique like FLAWS, focusing on the grey matter by attenuating the white matter and CSF signal. Finally, QSM sequences will be performed. QSM measures tissue magnetic susceptibility mostly influenced by iron, myelin and calcium content in the brain. Due to physical properties of the technique (bipolarity), we suppose that high resolution QSM will be more sensitive that previous used sequences to depict cortical lesions. Using this multi-contrast approach with relevant MRI sequence and with a high resolution whole brain exploration might improve the detection of CL in early MS.

Furthermore, MRI protocol allow us to estimate neuronal loss (T1 relaxation time), myelin and iron content (QSM and T2* relaxation time) within and outside cortical lesions in GM.

The present study is an opportunity to assess cortical pathology in MS from the onset of the disease, allowing to a better understanding of its origins and its impact and disease severity. This study is a preliminary requirement to longitudinal studies to precisely depict the kinetic of cortical lesion accumulation and the links with disease aggravation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting MS (McDonald's criteria 2010) early (duration evolution <2 years),
* Age between 18 and 45 years,
* No history of neurological symptoms suggestive of demyelinating pathology,
* No corticosteroids in the month preceding the completion of the MRI,
* Realization of the MRI in the first 6 months following the inaugural clinical episod

Exclusion Criteria:

* Argument for a differential diagnosis (systemic lupus erythematosus, antiphospholipid syndrome, Behçet's disease, sarcoidosis, Lyme disease, cerebral arteritis, lymphoma CNS, etc.),
* History of neurological or psychiatric illness,
* History of taking immunosuppressive drugs,
* Claustrophobia
* Pregnancy,
* Patient unable or unwilling to give consent, patient under guardianship,
* Patient not affiliated to a social security regime

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
visualization of cortical lesions | 12 MONTHS
  By IRM 7T

SECONDARY OUTCOMES:
measure of physical disability | 12 months
  score EDSS
cognitive impairment index | 12 months
  score IAC

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France